CLINICAL TRIAL: NCT02724033
Title: Comparative Study of Superficial Cervical Plexus Block and Nerve of Arnold Block With Intravenous Antiemetic Drugs Dexamethasone and Ondansetron and Incidence of Post-operative Nausea Vomiting for Inner Ear Surgery
Brief Title: Comparative Study of Superficial Cervical Plexus Block and Nerve of Arnold Block and Incidence of PONV for Inner Ear Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI has left Riley Anesthesia. Lack of staff for continued recruitment
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Charles W. Yates, MD, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Inner Ear PONV_Nouri
Record Dates: First submitted 2015-04-21; First posted 2016-03-31 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-05

CONDITIONS: Anesthesia, Pediatrics, Surgery
Keywords: post operative nausea vomiting; Inner ear surgery
MeSH Terms: interventions — Bupivacaine; Antiemetics; Dexamethasone; Calcium Dobesilate; Ondansetron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator): Group A - regional nerve block
  Interventions: Procedure: regional nerve block
- Group B (Active Comparator): Group B - antiemetic
  Interventions: Drug: Antiemetic
- Group C (Active Comparator): Group C - block and antiemetic
  Interventions: Procedure: regional nerve block; Drug: Antiemetic

INTERVENTIONS:
Procedure: regional nerve block — regional nerve block
  Other Names: Bupivacaine
  Arms: Group A; Group C
Drug: Antiemetic — Antiemetic
  Other Names: Dexamethasone (Decadron); ondansetron (Zofran)
  Arms: Group B; Group C

SUMMARY:
The investigators would like to compare the therapeutic and cost effectiveness of established therapies for postoperative nausea and vomiting to regional nerve blocks of the head and neck area an intervention known for analgesia but for which the antiemetic effects hasn't been entirely explored.

The rational is based on the knowledge of the anatomical innervation of the inner ear and the role of the parasympathetic nervous system in the emetic act. A lot of focus has been given on its counterpart the sympathetic nervous system and its role in painful conditions. The investigators believe that the nerve blockade of the parasympathetic innervation can have some beneficial effect in the post-surgical patient.

DETAILED DESCRIPTION:
The researchers hypothesize another potential antiemetic mechanism by the blockade of the auricular branch of the vagus nerve at the ear canal (commonly described as nerve of Arnold) in conjunction with a block of the greater auricular nerve and lesser occipital nerve at the superficial cervical plexus level. The block would cover both the sensory innervation and of the ear canal and the inner ear. A regional anesthetic block prior to the surgical intervention on the inner ear at the superficial cervical plexus block is performed. This latter is a branch of the vagus nerve at the superficial cervical plexus (erb's point). The block would inhibit the vagal afferent to area postrema through inhibition of afferent vagal input to the medullary center.

The emetic act (vomiting) is a highly integrated physiologic reflex involving both the somatic and autonomic nervous system. Researchers do not know how much of a relation there is between the vagal nerve branches involvement and incidence of nausea and vomiting effects are from the inner ear injury and or the inflammatory response type of response triggering the area postrema. The usual prophylactic treatment of PONV (post operative nausea and vomiting) has been limited to anti-emetics such as dexamethasone along with aggressive fluid therapy and adequate analgesia.

Investigators are proposing to conduct a comparative study of the therapeutic and cost effectiveness of regional anesthesia and antiemetic therapy in the prevention and treatment of PONV in children undergoing inner ear surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patient Age 1-18 yo
* Scheduled to have cochlear implantation, Tympanomastoidectomy, inner ear surgery
* Past history of PONV susceptibility

Exclusion Criteria:

* Patient/ Parents refusal
* Infection at the site of local anesthetic injection
* Known coagulopathy
* Existing VP shunt
* Severe mental disability
* Any known allergic to dexamethasone (Decadron) and/or ondansetron ( Zofran)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malik Nouri, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 11 | 14 | 12
Completed | 11 | 14 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 11 | 14 | 12 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 14 | 12 | 37
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8 | 16
  Male | 8 | 9 | 4 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11 | 14 | 12 | 37
Nausea [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0
Retching [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0
Nausea and Retching [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Post Operative Nausea and Vomiting
Description: number of patients with evidence of post operative nausea and vomiting
Time Frame: Post Operative within 24 hour Follow up Period
Population: Patients that had inner ear surgery and the above randomized intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 11 | 14 | 12
Participants
  Nausea | 6 | 6 | 4
  No Nausea | 5 | 8 | 8

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 1/11 | 1/14 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=11) | Group B (N=14) | Group C (N=12)
Hives (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Number of patients is less than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT02724033/Prot_SAP_000.pdf